CLINICAL TRIAL: NCT06436222
Title: Effectiveness of High Velocity Nasal Insufflation (HVNI) in Infants <32 Weeks Gestational Age(GA) or Birth Weight <1500 Grams With Moderate Respiratory Distress in Dr.Cipto Mangunkusumo Hospital
Brief Title: Effectiveness of HVNI in Preterm Infants With Moderate Respiratory Distress
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Putri Maharani Tristanita Marsubrin, Sp. A(K), Principal Investigator of Perinatology Division, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 336/UN2.F1/ETIK/PPM.00.02/2024
Record Dates: First submitted 2024-05-20; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Distress, Newborn
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups either HVNI (intervention group) or CPAP (control group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HVNI (Intervention Group) (Other): The infant was given therapy using HVNI with an initial flow of 6 L/min. Inspiratory fraction of oxygen (FiO2) started with 30% following the SpO2 target. The maximum flow is 8L/min. FiO2 can be increased by 5% until the target SpO2 is reached.
  Interventions: Device: HVNI
- CPAP(Control Group) (Other): The infant was given therapy using CPAP with an initial pressure of 7 cmH20. Inspiratory fraction of oxygen (FiO2) starting with 30% following the SpO2 target.The maximum of CPAP pressure is 8 cmH2O. FiO2 can be increased by 5% until the target SpO2 is reached.
  Interventions: Device: HVNI

INTERVENTIONS:
Device: HVNI — Preterm infants with gestational age (GA) less than 32 weeks or birth weight less than 1500 grams. The infant has moderate respiratory distress (Downe score ≤ 6) detected within 24 hours after birth.

SUMMARY:
Neonatal respiratory distress is a common problem in preterm infants. The application of CPAP is widely used in neonatal units as a primary mode of respiratory support for respiratory distress. However, discomfort, nasal injuries, and fixation difficulties have been reported as obstacles when applying CPAP. High velocity nasal insufflation (HVNI) may serve as an alternative to CPAP. Trials are needed to evaluate the effectiveness of HVNI in reducing the incidence of respiratory distress. The aim of this study is to compare the clinical effectiveness and safety of HVNI as an alternative therapy to CPAP in premature infants with moderate respiratory distress. This study is a prospective, non-inferiority, randomized, unblinded controlled trial to compare the efficacy of HVNI and CPAP. The subjects were randomly allocated to receive either HVNI or CPAP according to the study protocol. They were randomly assigned using blocks of four. The completion of HVNI therapy was determined by therapeutic failure within 72 hours following enrollment, indicated by the need for intubation.

ELIGIBILITY:
**Inclusion Criteria:**

* Preterm infants born in Cipto Mangunkusumo Hospital with gestational age (GA) less than 32 weeks or birth weight less than 1500 grams.
* Infants with moderate respiratory distress (Downe score ≤ 6) detected within 24 hours after birth.
* Parents are willing to participate in the study.

**Exclusion Criteria:**

* Infants with severe respiratory distress (Downe score ≥ 6) requiring invasive treatment in the form of mechanical ventilation, or apnea indicated by surfactant administration via endotracheal tube.
* Infants with contraindications to the use of non-invasive ventilation such as esophageal atresia, diaphragmatic hernia, air leak syndrome, and other conditions.
* Infants with respiratory distress due to non-pulmonary abnormalities.
* Infants with congenital metabolic disorders.
* Infants with congenital abnormalities that exacerbate respiratory distress.

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of HVNI to prevent intubation within 72 hours | Intubation rates within 72 hours
  The primary outcome was treatment failure/success within 72 hours of treatment between HVNI and CPAP

SECONDARY OUTCOMES:
Length of stay | 30 days
  Duration from birth until discharge

OTHER OUTCOMES:
Intraventricular Hemmorhage (IVH) | one week
  The occurrence of bleeding in lateral and third or fourth ventricles characterized by hyper-attenuating fluid typically seen as layering within the ventricles in imaging studies
Bronchopulmonary Dysplasia (BPD) | Within 28 days
  Prolonged need for supplemental oxygen in preterm infants after 28 days of age or after 36 weeks postmenstrual age and who do not have other conditions requiring oxygen

IPD SHARING:
Plan to Share IPD: No